CLINICAL TRIAL: NCT00093860
Title: Propranolol for Syncope With Sympathoadrenal Imbalance in Children
Brief Title: Propranolol to Treat Fainting in Children With Sympathoadrenal Imbalance
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 050001; 05-N-0001
Record Dates: First submitted 2004-10-06; First posted 2004-10-07 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-03

CONDITIONS: Syncope
Keywords: Adrenaline; Norepinephrine; Sympathetic Nervous System; Fainting; Hypotension; Beta-Adrenoceptors; Neurocardiogenic Syncope; Chronic Orthostatic Intolerance; Sympathoadrenal Imbalance; SAI; Children
MeSH Terms: conditions — Syncope; Hypotension; Syncope, Vasovagal | interventions — Propranolol

INTERVENTIONS:
Drug: Propranolol

SUMMARY:
This study will examine the effectiveness of the drug propranolol in preventing fainting in patients with sympathoadrenal imbalance (SAI). SAI is a particular pattern of nervous system and chemical responses in which the blood vessels in skeletal muscles do not remain constricted appropriately during standing for a long time. This can lower blood pressure and cause fainting. Propranolol (Inderal® (Registered Trademark)) is a Food and Drug Administration-approved drug that belongs to a class of drugs called beta-blockers. These drugs slow the heart rate and maintain blood pressure in certain situations.

Children between 10 and 17 years of age with frequent fainting or near-fainting due to SAI may be eligible for this study. Children must experience severe dizzy episodes at least once every 2 months or fainting episodes at least once every 4 months. The condition must be severe enough to affect the child's quality of life or to have forced the child to alter his or her life routines to accommodate to the illness. Screening includes a tilt table test, described below, to determine if the child has a particular chemical pattern in the blood.

Children enrolled in the study take propranolol pills in increasing doses during the first week of the study to determine the proper dose for the individual. Then, the drug is stopped until the experimental phase of the study begins. In this phase, children are randomly assigned to take either propranolol or placebo (a look-alike pill with no active ingredient) for a maximum of 3 days. On the fourth day, the child undergoes a tilt table test to determine whether the treatment affects his or her ability to tolerate tilt. For this test, the child lies on a padded table with a motorized tilt mechanism that can move the child from a flat position to an upright position in about 10 seconds. The child remains upright for up to 40 minutes while the following measurements are taken:

* Blood sampling: Blood is drawn through a catheter (thin plastic tube) placed in an arm vein. This allows repeated sampling without repeated needle sticks. Samples are collected before starting the tilt test, about every 4 minutes during the test, immediately when a drop in blood pressure is detected or symptoms develop, and after 10 minutes of recovery lying flat. A maximum of 12 samples are collected for each tilt test.
* Physiologic measurements: Blood pressure, heart rate, and electrocardiogram (EKG) are measured continuously during the tilt test session, and blood flows and skin electrical conduction are measured intermittently. Blood flow is measured using sensors applied to the skin and a blood pressure cuff around the limb. For skin blood flow measurements, a laser beam scans the skin surface. The skin electrical conduction test measures how well the skin conducts electricity. This is measured through sensors placed on the tips of two fingers. Respiration and breathing rate are monitored by an elastic cloth band around the chest.
* Self-report questionnaires: Patients or their parents complete a questionnaire about the child's symptoms before and during treatment.

The effects of the test drug are allowed to wear off for up to 1 week, after which the entire tilt test procedure is repeated. Patients who were given propranolol for the first test session take placebo for the repeat session, and those who were given placebo take propranolol.

DETAILED DESCRIPTION:
Objectives: This protocol is to evaluate treatment with oral propranolol for a particular form of neurocardiogenic syncope (NCS), characterized by a neuroendocrine pattern called "sympathoadrenal imbalance" (SAI), in children. In SAI, plasma adrenaline levels increase progressively and to a greater extent than do norepinephrine levels, before syncope. The SAI pattern is associated with skeletal muscle vasodilation. We hypothesize that increased occupation of beta-2 adrenoceptors in skeletal muscle by high circulating adrenaline levels precipitates the neurocirculatory positive feedback loop that leads to NCS.

Study Population: Patients 10-17 years old with a history of NCS.

Design: In a randomized, crossover-design, placebo-controlled, double-blind trial, we test the above hypothesis by using the non-selective beta-adrenoceptor blocker, propranolol. We predict that in patients with previously documented SAI and tilt-evoked NCS, propranolol treatment will improve orthostatic tolerance during follow-up tilt table testing.

Outcome Measures: The primary outcome measure will be whether propranolol therapy can prevent tilt induced syncope; or significant hypotension and/or bradycardia preceding development of clinical symptoms (greater than or equal to 20 mm Hg decrease in blood pressure or heart rate less than 40 beats/min). Secondary dependent measures that will be assessed are occurrence of duration of tilt tolerance (if tilt induced symptoms are provoked), hemodynamic and neurochemical indices of SAI, and patient questionnaire reports.

ELIGIBILITY:
INCLUSION CRITERIA:

Subjects are patients referred for evaluation of chronic orthostatic intolerance. Patients enter into the therapeutic trial after they are determined to have NCS with SAI in a screening evaluation. Participation in this protocol is offered to individuals 10-17 years of age, independently of gender, race, ethnicity, religion, or any other demographic or sociopolitical classifications. To be eligible to enter this study, the patient must have a minimum frequency of pre-syncope of at least 1 event/2 months, or syncope of at least once/4 months. The severity of the symptoms should be of such severity as to alter the individual's quality of life or routines of life.

EXCLUSION CRITERIA:

Age: Minors younger than 10 years old and pregnant female subjects between 10 and 17 years of age will be excluded.

Risk: A candidate subject is excluded if, in the judgment of the Principal Investigator, protocol participation would place the subject at substantially increased acute medical risk. This includes the risk associated with air travel to the NIH. A candidate subject is excluded if, in the opinion of the Principal Investigator, the medical risk outweighs the potential scientific benefit.

Disqualifying Conditions: A candidate subject is excluded if there is a disqualifying condition. Examples of disqualifying conditions are history of asthma or chronic obstructive pulmonary disease requiring bronchodilators, hepatic or renal failure, atrioventricular block of any degree, bradycardia, symptomatic congestive heart failure, severe anemia, psychosis, refractory ventricular arrhythmias, insulin-dependent diabetes mellitus, or psychiatric disorders requiring continuous drug treatment. Patients with known allergy or hypersensitivity to propranolol are excluded from this study. A positive HIV test result does not necessarily exclude a patient from participating. If a female subject becomes pregnant during the study, she will be excluded from further participation in the study.

Medications: A candidate subject is excluded if clinical considerations require that the patient continue treatment with a drug likely to interfere with the scientific results. Patients who must take medications daily in the following categories are excluded: anticoagulants, tricyclic antidepressants, barbiturates, aspirin, acetaminophen, insulin, and bronchodilators. Patients are not to discontinue any medications before the patient or the patient's doctor discusses this with the Principal Investigator, an Associated Investigator, or Research Nurse. If it is decided that discontinuing medications would be unsafe, then the patient is excluded from the study.

Herbal Medicines and Dietary Supplements: Certain herbal medicines or dietary supplements are known or suspected to interfere with the experimental results, and such herbal medicines or dietary supplements must be discontinued before enrollment in the study. For many herbal medicines or dietary supplements, the mechanisms of action and therefore the possible effects on the experimental results are unknown. In cases where the subjects wish to continue their herbal medicines or dietary supplements while in study, and search the available medical literature fails to identify effects that are known or expected to interfere with the experimental results, then the subjects may participate.

Practical Limitations: Patients in whom we feel it would be difficult to technically carry out the testing procedures are excluded.

Pregnancy: Pregnant or lactating females of child-bearing potential are excluded. A blood test pregnancy will be conducted in all females of childbearing potential, before intake evaluation and also before each drug treatment phase. During the course of the protocol, patients who are of childbearing potential will be advised to practice adequate contraception (birth control pills, Depo-Provera, or implanted intrauterine device), if sexually active. If during the course of this study, a minor patient is found to have a positive pregnancy test, she will be asked confidentially whether she has had any recent sexual activity that could have resulted in the test being positive. In agreement with current legal statutes, the minor patient will be told confidentially that she is pregnant. She will be encouraged to share this information with her parents. By current legal statutes, we will not directly divulge this information to her parents. The pregnant minor subject will also be told that further participation in the study is a protocol violation (because of possible adverse risks to the unborn fetus), and she will be terminated from continued participation in the protocol.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50
Dates: Start 2004-10; Study Completion 2005-03

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Robertson RM, Medina E, Shah N, Furlan R, Mosqueda-Garcia R. Neurally mediated syncope: pathophysiology and implications for treatment. Am J Med Sci. 1999 Feb;317(2):102-9. doi: 10.1097/00000441-199902000-00004. PMID 10037113
- [Background] Goldstein DS, Holmes C, Frank SM, Dendi R, Cannon RO 3rd, Sharabi Y, Esler MD, Eisenhofer G. Cardiac sympathetic dysautonomia in chronic orthostatic intolerance syndromes. Circulation. 2002 Oct 29;106(18):2358-65. doi: 10.1161/01.cir.0000036015.54619.b6. PMID 12403667
- [Background] Jacobs MC, Goldstein DS, Willemsen JJ, Smits P, Thien T, Dionne RA, Lenders JW. Neurohumoral antecedents of vasodepressor reactions. Eur J Clin Invest. 1995 Oct;25(10):754-61. doi: 10.1111/j.1365-2362.1995.tb01954.x. PMID 8557062